CLINICAL TRIAL: NCT00838487
Title: Phase 3 Study, to Evaluate Safety & Efficacy of the Association Condroflex + Therapeutic Exercises Compared to Placebo + Therapeutic Exercises, in Subjects With Knee OA
Brief Title: Evaluate Safety & Efficacy of Condroflex in Subjects With OA
Acronym: ZD20108
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zodiac Produtos Farmaceuticos S.A. (Industry)
Responsible Party: Julio Cesar Nophal de Carvalho, Zodiac Produtos Farmaceuticos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZODIAC
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Treatment; Osteoarthritis; Elderly
Keywords: chondroitin; glucosamine; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- condroflex and exercise (Active Comparator): assent arm
  Interventions: Other: condroflex and exercise
- sugar pill and exercise (Placebo Comparator): sugar pill arm
  Interventions: Other: sugar pill and exercise

INTERVENTIONS:
Other: condroflex and exercise — 1 sachet oral once a day by 12 Weeks / therapeutic exercise 3 times a week
  Other Names: glucosamine sulph + chondroitin sulph and therapeutic exerc.
  Arms: condroflex and exercise
Other: sugar pill and exercise — 1 sachet oral once a day by 12 Weeks / therapeutic exercise 3 times a week
  Other Names: Placebo Comparator and therapeutic exerc.
  Arms: sugar pill and exercise

SUMMARY:
Primary Objective: To compare, after 12 weeks of double-blind treatment, the evolution of the improvement of pain (at rest and during / after exercise) in the questionnaire WOMAC (Western Ontario and McMaster Universities Arthritis Index), achieved with Condroflex ® oral administration(sulfate glucosamine + chondroitin sulfate sodium) in association with therapeutic exercises, compared to placebo in association with therapeutic exercises in individuals with knee OA and not exposed to prior treatment with the products under investigation.

DETAILED DESCRIPTION:
To have osteoarthritis degree 2 or 3 / To be capable to consent

ELIGIBILITY:
Inclusion Criteria:

* to have knee osteoarthritis degree 2 or 3
* to be capable to consent

Exclusion Criteria:

* previous drug treatment
* concomitant diseases
* concomitant drugs

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-07 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
improvement of pain | 12 week

SECONDARY OUTCOMES:
rigidity restriction | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Suely Roizenblatt, Principal Investigator — CRM Regional Council of Medicine
Locations (1):
- CRDB, São Paulo, Brazil